CLINICAL TRIAL: NCT05333991
Title: Endothelial Leakage Assessed by 125-I Labeled Serum Albumin and the Association to Endothelial Biomarkers After Major Abdominal Surgery
Brief Title: Endothelial Leakage and the Association to Endothelial Biomarkers After Surgery
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sandra Taylor Pitter, clinical professor, Rigshospitalet, Denmark
Other Study IDs: 2022-RH-iod-tracer
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Pancreas Disease
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Plasma is collected from blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of this study is to investigate fluid loss from the blood stream (''endothelial leakage'') and the damage on the vessel wall (''endothelial function'') during surgery.

Cardiovascular complications during surgery are said to have different causes, e.g. lack of fluid in the blood stream (''hypovolemia'') and decreased vascular tone. Hypovolemia can have different causes, one being damage to the endothelial function. During trauma and infection, it has been previously shown, that damage to the endothelial function causes fluid loss from the blood stream. Nevertheless, this has never been demonstrated during surgery.

Secondary this study will measure the blood flow using a thermo-camera during surgery. This will together with selected blood tests provide information on various possible causes to hypovolemia.

The purpose of this study is to describe and quantify endothelial damage (assessed by selected endothelial biomarkers) and albumin escape rate as a proxy for endothelial leakage (assessed by measuring radioactive 125-I labeled HSA injected postoperatively), combined with assessment of MTS (assessed by Laser Speckle Contrast Imaging (LSCI) and digital thermography). This will allow a detailed description of the surgery's impact on the endothelial integrity and contribute to a better understanding of the physiological changes that occur postoperatively.

The study will investigate patients undergoing pancreaticoduodenectomy (Whipple) and total pancreatectomy. These patients have a vast clinical need, being one of the most extensive abdominal surgical procedures with great stress response.

The study is a prospective exploratory cohort study and methods include blood sampling pre- and post-operatively, 125-I labeled humane serum albumin postoperatively (and preoperatively if logistically possible) and thermography.

The hypothesis of this study is that the extent of endothelial damage measured by selected biomarkers is associated with the level of albumin escape rate after major abdominal surgery. Secondly, inflammation increases albumin escape rate after major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients are scheduled for Whipple or total pancreatectomy

Exclusion Criteria:

* Patient having received immunomodulating treatments less than four weeks prior to surgery
* Patient having other major surgery performed less than four weeks prior to surgery. Thus, minor surgery allowed, for instance minor skin incisions
* Patient having endoscopic retrograde cholangiopancreatography (ERCP) or Percutaneous transhepatic cholangiography (PTC) performed less than two weeks prior to surgery
* Patients scheduled for major vascular surgery during Whipple or total pancreatectomy
* Patient is diagnosed with chronic kidney failure or is in diuretics treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major abdominal surgery patients will be included. Patients are screened prior to surgery from electronic medical charts. Patients can be co-enrolled in other non-intervention trials. An outline of scheduled study activities is shown in figure one.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Albumin escape rate during the first five postoperative days assessed by intravascular loss of 125-I labeled HSA. | five days after surgery
  Measured by the use of iod tracer

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The data for all included patients will be available for other selected research colleagues
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Up to 5 years after data collected